CLINICAL TRIAL: NCT05017714
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy of Aerosolized Novaferon in Asymptomatic and Mildly Symptomatic Patients Infected With SARS-CoV-2.
Brief Title: A Trial of Novaferon in Asymptomatic or Mild COVID-19 Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Jing302H
Record Dates: First submitted 2021-08-18; First posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: SARS-CoV2 Infection
MeSH Terms: conditions — COVID-19 | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active plus SOC (Experimental)
  Interventions: Drug: Recombinant cytokine gene derived protein injection
- Placebo plus SOC (Placebo Comparator)
  Interventions: Drug: Recombinant cytokine gene derived protein injection

INTERVENTIONS:
Drug: Recombinant cytokine gene derived protein injection — Aerosolized Novaferon, given 20 ug BID, daily for 7 days, plus Standard of Care.
  Inhaled Saline (placebo), given BID, daily for 7 days, plus Standard of Care.
  Other Names: Saline

SUMMARY:
This is a phase III randomized, double blinded, placebo-controlled multi-center study to assess the efficacy and safety of aerosolized Novaferon for the treatment of asymptomatic or mildly patients infected with SARS-CoV-2.

DETAILED DESCRIPTION:
Since the outbreak of New Coronavirus pneumonia (COVID-19) in late 2019, epidemics around the world are still developing. There are about 200 million confirmed cases in the world, including about 4.26 million deaths until August 5, 2021, which has become a major disaster for human being.

Most of SARS-CoV-2 infection are asymptomatic or mild cases, which is the main factor causing viral transmission. Although COVID-19 patients have immune protection after cured or vaccinated, there still be a percentage of people vaccinated who still get sick, hospitalized, or die caused by COVID-19. COVID-19 vaccine breakthrough and reinfection cases became one of key problems for COVID-19 prevention and control. In addition, SARS-CoV-2 variants circulated in the world. However, some variants were associated with disease severity, the performance of vaccines, therapeutic medicines, diagnostic tools, or other public health and social measures. Variants (e.g., Delta variant) caused some vaccine breakthrough cases. There is an urgent need for effective antiviral drugs.

Novaferon is a marketed antiviral drug in China and proved to have more than ten-fold antiviral potency than that of similar interferon α-2b. Novaferon exerts antiviral activity by three ways: blocking virus entry into cells, inducing expression of antiviral genes and proteins (e.g., MX1 and OAS), and promoting apoptosis of infected cells. In vitro experimental study showed Novaferon exhibited anti-SARS-CoV-2 effects at the cellular level. A randomized, open-label, parallel-group trial demonstrated that aerosolized Novaferon expedited clearance and negative conversion of SARS-CoV-2, which provide the rational for large-scale clinical studies to verify the efficacy of Novaferon as a potential antiviral drug for COVID-19. Inhalation administration has advantages over systemic administration in reducing adverse drug reactions, promoting the distribution of drugs in respiratory tract, and thus enhancing the mucosal immunity.

This is a phase III randomized, double blinded, placebo-controlled multi-center study to assess the efficacy, and safety of aerosolized Novaferon for the treatment of asymptomatic patients or patients with mild COVID-19.

ELIGIBILITY:
Inclusion Criteria:1.Patient capable of giving consent, or, when the patient is not capable of giving consent, by his or her legal/authorized representatives prior to initiation of any study procedures.

2.Male or female, between 18 and 65 years of age at the time of consent. 3.Laboratory-confirmed SARS-CoV-2 infection as determined by RT-PCR in nasopharyngeal or oropharyngeal swabs < 72 hours prior to enrollment.

4Patients with asymptomatics or mild COVID-19, including:

1. Patients with asymptomatic infections refer to those with positive testing results in etiological detection of SARS-CoV-2 in swabs, but without any relevant clinical manifestations, such as self-perceived or clinically identified symptoms or signs, including fever, cough and sore throat, and without any typical imaging features of COVID-19 in their CT scans.
2. Patients with mild SARS-COV-2 infections refer to those who are infected with SARS-COV-2 presenting mild symptoms in accordance with Diagnosis and Treatment Protocol for Novel Coronavirus Pneumonia (Trial Revision 8): mild clinical symptoms, and no findings of pneumonia in chest CT images.

   -

Exclusion Criteria:1.Patients classified into Moderate, Severe, and Critical cases according to the Diagnosis and Treatment Protocol for Novel Coronavirus Pneumonia (Trial 8th Edition) 2.Females who are breast-feeding, lactating, pregnant or intending to become pregnant 3.Patients who are receiving any treatment with interferon or participating in other clinical studies of antiviral therapy.

4.Patients who are unable to collaborate due to poor mental health, suffering from psychiatric illness, or incapable of controlling themselves or expressing clearly.

5.Patients excluded in the opinion of the investigators.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-08-31 (Estimated); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Time of negative detection of SARS-CoV-2 RNA | Day 1 to Day 28
  Nucleic acid detection twice at a 24-hour interval

SECONDARY OUTCOMES:
Rate of clinical progression | Day 1 to Day 28
  at least 4 points on 8-point ordinal Scale developed by WHO
the change of viral load | Day 1 to Day 28
  viral load cannot be detected
detection rate of SARS-CoV-2 RNA | Day 1 to Day 28
  cannot detect SARS-CoV-2 RNA
Rate of clinical progression in patients vaccinated | Day 1 to Day 28
  Time of negative detection of SARS-CoV-2 RNA in patients vaccinated
Rate of clinical progression in subgroup of patients vaccinated | Day 1 to Day 28
  at least 4 points on 8-point ordinal Scale developed by WHO
Rate of clinical progression in patients infected with variants( Delta strain, et al) | Day 1 to Day 28
  at least 4 points on 8-point ordinal Scale developed by WHO
Safety and tolerability | Day 1 to Day 28
  AE score